CLINICAL TRIAL: NCT04705012
Title: SPiT-frequency; the Effect of Increased Frequency of Intervention, Using Chitosan Brushes, on Post-surgical Peri-implant Inflammation
Brief Title: SPiT-frequency; the Effect of Increased Frequency of Intervention on Post-surgical Peri-implant Inflammation
Acronym: SPiT-freqvzy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Odd Carsten Koldsland, Associate professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 195347
Record Dates: First submitted 2020-12-17; First posted 2021-01-12 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Peri-Implantitis
Keywords: SPiT
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Examiner blinded split-mouth clinical trial
Who Masked: Outcomes Assessor
Masking Description: The assessor will not participate in the treatment, is blinded to what implant receives which treatment and leaves the room following examination prior to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - increased frequency of submucosal cleaning (Experimental): At follow-up time points (3-, 6-, 9-, 16 weeks) following initial treatment), all implants receive supramucosal polishing, but only test-implants receive submucosal debridement 12 + 24 +36 weeks following baseline: all implants receive supramucosal polishing as well as submucosal debridement as described above
  Interventions: Other: Submucosal supportive therapy
- Control - conventional frequency of submucosal cleaning (Active Comparator): At follow-up time points (3-, 6-, 9-, 16 weeks) following initial treatment), all implants receive supramucosal polishing, but only test-implants receive submucosal debridement 12 + 24 +36 weeks following baseline: all implants receive supramucosal polishing as well as submucosal debridement as described above
  Interventions: Other: Submucosal supportive therapy

INTERVENTIONS:
Other: Submucosal supportive therapy — Increased frequency of submucosal cleaning using a rotating chitosan brush

SUMMARY:
This pilot study is an interventional clinical study on the supportive peri-implant treatment (SPiT) necessary to maintain/ improve the clinical conditions surrounding a dental implant following surgical treatment of peri-implantitis. The focus of this pilot, double arm, split-mouth, single centre, controlled, randomised clinical study is to examine the effect of short-term increased frequency of a SPiT-protocol.

DETAILED DESCRIPTION:
Patients with surgically treated peri-implantitis enrolled in a maintenance program at the Specialist clinic, Institute for Clinical Dentistry, Dental Faculty, University of Oslo, will receive SPiT by the use of an oscillating chitosan brush (LBC, BioClean, Labrida AS, Oslo, Norway). Subjects with at least two not-adjacent implants of similar brand and defect configuration registered with suppuration or Bleeding index score 3-2 (Roos-Jansaker et al., 2007) on at least 1 of 6 surfaces (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) will be invited to participate in the current pilot study.

Baseline examinations and treatment:

Radiographs of the implants showing clear projections of the implant threads at the mesial and distal surfaces will be taken using standard Eggens holders

The following clinical registrations will be performed at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) of the included implants by the blinded examiner:

Suppuration: the presence or absence after light pressure against gingiva/mucosa or following gentle probing of the peri-implant pocket.

Plaque: the presence or absence recognized by running a probe across the marginal surface of the implant (Mombelli, van Oosten, Jr, & Lang, 1987).

Gingival bleeding: registered according to the Modified Sulcus Bleeding Index (mBI) (Mombelli et al., 1987).

PPD: recorded with a pressure- sensitive probe (20 g) (University of North Carolina probe, Aesculap, Braun, Tuttlingen, Germany).

Bleeding index score: measured at the implants after probing at six sites, and graded (0-3):

0 = no bleeding,

1. = spot bleeding,
2. = line bleeding
3. = profound bleeding within 30 seconds after measurement of PPD. Presence of keratinized mucosa: registered at the mid buccal site as "adequate" ≥2 mm, "inadequate" <2 mm (Moraschini, Luz, Velloso, & Barboza, 2017).

All included implants receive the following treatment:

Repeated oral hygiene instruction if needed Submucosal debridement with a chitosan brush (LBC, BioClean®, LABRIDA AS, Oslo, Norway) seated in an oscillating dental drill piece (ER10M, TEQ-Y, NSK Inc., Kanuma Tochigi, Japan) for 3 min followed by copious irrigation with sterile saline Supramucosal polishing using polishing paste and rubber cup Following treatment, if local anesthesia was not applied, the subjects will be asked to grade the level of pain experienced on a 10 cm visual analogue scale (VAS).

3-, 6- and 9 weeks following baseline At the 3-week follow up, an equal number of included implants are determined "test-" and "control-" by flipping of a coin.

At these time points, all implants are clinically examined by a blinded examiner and receive supramucosal polishing, but only test-implants receive submucosal debridement as described above (see figure 1) VAS scales are registered

12 weeks (3 month) following baseline At these time point, all implants are clinically examined by a blinded examiner and receive supramucosal polishing as well as submucosal debridement as described above (see figure 1) VAS scales are registered

16 weeks (4 month) following baseline All implants are clinically examined by a blinded examiner and receive supramucosal polishing, but only test-implants receive submucosal debridement as described above (see figure 1) VAS scales are registered

24 weeks (6 month) following baseline At these time point, all implants are clinically examined by a blinded examiner and receive supramucosal polishing as well as submucosal debridement as described above (see figure 1) VAS scales are registered

36 weeks (9 month) following baseline At these time point, all implants are clinically examined by a blinded examiner and receive supramucosal polishing as well as submucosal debridement as described above (see figure 1) VAS scales are registered Radiographs are taken according to the baseline examination

Figure 1: Timeline of the clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 20 years,
* Subjects must have received surgical treatment of peri-implantitis as defined by the World Workshop 2017 criteria (Berglundh et al., 2018).
* Subjects have to present inflammation (suppuration or BoP 3-2) at more than one implant of similar implant brand, with similar defect type (Schwarz et al., 2007), and defect severity.
* The implants must not be replacing adjacent teeth (minimum space for one tooth/implant between test and control.

Exclusion Criteria:

* • Previous radiotherapy in the affected area, current use of chemotherapy, systemic long-term corticosteroid treatment.

  * No pregnant or nursing subjects.
  * < class 2 according to the ASA (American Society of Anesthesiologists) physical status classification.
  * Registered implant bone loss with exposed modified surface < 2.0 mm.
  * If examiners/operators agree the placement of the implant (angle, position, proximity to adjacent implant or tooth) or suprastructure was suboptimal and considered to play a major role in the development and sustain the peri-implant disease.
  * Anatomical abnormalities
  * clinical exclusion criteria specific to the disease/condition
  * specific concomitant treatment with other devise, mouthrinse or systemic antibiotics
  * participation in any other clinical study within the last month
  * inability to comprehend and respond to the quality of life questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Eradication of disease | 9 months
  Proportion of implants without signs of inflammation defined as BoP and/or suppuration (eradication of disease)

SECONDARY OUTCOMES:
Reduction in inflammation, | 9 months
  changes in severity of inflammation (inflammation assessed as Bleeding index 3, 2 or 1 (Roos-Jansaker et al., 2007)
Radiographic changes | 9 months
  progressive bone loss as measured on radiographs
Morbidity, patient centered outcomes | 9 month
  patient experience of pain in relation to treatment
Implant survival | 9 month
  implant present at examination